CLINICAL TRIAL: NCT03863886
Title: Endoscopic Ultrasound Determines Disease Activity in Crohn's Disease And Ulcerative Colitis
Acronym: EUSIBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, Vu Nguyen, Assistant Professor of Medicine, Carilion Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2694
Record Dates: First submitted 2019-01-22; First posted 2019-03-05 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Crohn Disease; Ulcerative Colitis
Keywords: crohn's disease; ulcerative colitis; endoscopic ultrasound; inflammatory bowel disease
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Crohn's Disease (Experimental): 20 patients with Crohn's disease with at least colonic involvement will undergo endoscopic ultrasound assessment of the thickness of wall layers (mucosa, submucosa, muscularis propria, total wall) at the rectum and cecum region during their standard-of-care colonoscopy.
  Interventions: Procedure: Endoscopic ultrasound catheter (UM-2R/3R, Olympus)
- Ulcerative Colitis (Experimental): 20 patients with ulcerative colitis will undergo endoscopic ultrasound assessment of the thickness of wall layers (mucosa, submucosa, muscularis propria, total wall) at the rectum and cecum region during their standard-of-care colonoscopy.
  Interventions: Procedure: Endoscopic ultrasound catheter (UM-2R/3R, Olympus)
- Non-IBD Controls (Experimental): 20 patients without inflammatory bowel disease (controls) will undergo endoscopic ultrasound assessment of the thickness of wall layers (mucosa, submucosa, muscularis propria, total wall) at the rectum and cecum region during their standard-of-care colonoscopy.
  Interventions: Procedure: Endoscopic ultrasound catheter (UM-2R/3R, Olympus)

INTERVENTIONS:
Procedure: Endoscopic ultrasound catheter (UM-2R/3R, Olympus) — A miniprobe ultrasound catheter (UM-2R/3R, Olympus) will be passed into the colonoscope's accessory channel at the time of colonoscopy to measure the thickness of the different colon wall layers (mucosa, submucosa, muscular propria, and total wall thickness) in the cecum and rectum.

SUMMARY:
Although Crohn's disease and ulcerative colitis are the main subtypes of inflammatory bowel disease, they differ substantially in disease behavior, prognosis, and treatment paradigm. However, making an accurate diagnosis of Crohn's disease versus ulcerative colitis and assessing disease activity beyond the level of mucosal inflammation remain challenging with contemporary modalities. The objective of the study is to determine the novel role of endoscopic ultrasound in A) differentiating Crohn's colitis versus ulcerative colitis and B) monitoring disease activity in these patients.

DETAILED DESCRIPTION:
Crohn's disease (CD) and ulcerative colitis (UC) are two principal subtypes of inflammatory bowel disease (IBD). Disease behavior, prognosis, and therapy differ substantially between these two subtypes. However, up to 15% of patients may have misclassification of their IBD subtypes leading to significant delay in appropriate management and prognostication. The misclassification of CD and UC is due to limitations in contemporary modalities used to diagnose these diseases. While CD involves transmural inflammation and UC is limited to mucosal inflammation, the combination of endoscopy, histology, and cross-sectional imaging typically used to establish the diagnosis do not reliably distinguish mucosal from submucosal inflammation. Consequently, disease reclassification often occurs at the time of surgery when transmural inflammation can be determined from the surgical specimen. At that time, medical therapy has already failed. The optimal time for accurate IBD classification would be at the initial diagnosis, allowing for appropriate targeted therapy to achieve optimal disease outcomes.

Endoscopic ultrasound (EUS) can provide detailed information about luminal wall layers. To date, the use of endoscopic ultrasound (EUS) for colorectal disease has been limited to staging of subepithelial lesions and examining CD-related perianal complications. The ultrasound miniprobe device (UM-2/3R, Olympus) is a thin ultrasound catheter that can be passed through the colonoscope's accessory channel to perform detailed ultrasonic assessment of any colon wall segments. Prior studies have demonstrated that the submucosal layer is significant thicker in active CD compared to active UC, while active UC has thicker mucosal layer comparatively. This study tests the hypothesis that the addition of the miniprobe ultrasound catheter at the time of colonoscopy will help to differentiate active CD with colonic involvement and UC from non-IBD controls by comparing the differential thickness in the mucosal and submucosal layer among these groups of patients. Furthermore, the investigators hypothesize that the thickness of differential wall layers in CD and UC patients will correlate to clinical and endoscopic disease activity. The significance of these findings will help establish an accurate diagnosis of IBD subtypes early in the disease course and provide for a reliable method to monitor disease activity not only at the mucosal layer but also in deeper luminal wall layers.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients ≥ 18 years of age with CD with at least colonic involvement, UC, or non-IBD controls who have been referred for colonoscopy for clinical reasons. The clinical reasons may include colorectal cancer screening, surveillance, diagnostic for CD or UC flare, or gastrointestinal symptoms.

Exclusion Criteria:

* Pregnant patients.
* Patients with known current colorectal cancer, infectious colitis, diverticulitis, or microscopic colitis.
* Patients who have undergone surgery involving the cecum or rectum.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-04 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Active Crohn's disease has significantly thicker submucosa layer compared to patients with active ulcerative colitis and non-inflammatory bowel disease controls. | Day 1
  We are measuring the different colon wall layer thickness including the mucosa, submucosa, muscularis propria, and total wall layer (in mm) using the endoscopic ultrasound device and comparing the different levels of colon wall layer thickness between patients with active versus inactive ulcerative colitis, active versus inactive Crohn's disease, and comparing those to controls.

SECONDARY OUTCOMES:
The thickness of the submucosa layer in Crohn's disease patients correlates to the degree of disease activity as measured by the Harvey-Bradshaw clinical index and Simple Endoscopic Score index. | Day 1
  We will correlate the thickness (in mm) of the submucosa layer in Crohn's disease patients measured by endoscopic ultrasound to the degree of disease activity at the time of procedure as measured by the Harvey-Brashaw index and Simple Endoscopic Score (SES-CD) index.
The thickness of the mucosa layer in ulcerative colitis patients correlates to the degree of disease activity as measured by the Mayo score index. | Day 1
  We will correlate the thickness (in mm) of the mucosa layer in ulcerative colitis patients measured by endoscopic ultrasound to the degree of disease activity at the time of procedure as measured by the Mayo score index.

CONTACTS AND LOCATIONS:
Overall Officials: Vu Q Nguyen, M.D., Principal Investigator — Assistant Professor of Medicine
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gomollon F, Dignass A, Annese V, Tilg H, Van Assche G, Lindsay JO, Peyrin-Biroulet L, Cullen GJ, Daperno M, Kucharzik T, Rieder F, Almer S, Armuzzi A, Harbord M, Langhorst J, Sans M, Chowers Y, Fiorino G, Juillerat P, Mantzaris GJ, Rizzello F, Vavricka S, Gionchetti P; ECCO. 3rd European Evidence-based Consensus on the Diagnosis and Management of Crohn's Disease 2016: Part 1: Diagnosis and Medical Management. J Crohns Colitis. 2017 Jan;11(1):3-25. doi: 10.1093/ecco-jcc/jjw168. Epub 2016 Sep 22. PMID 27660341
- [Result] Magro F, Gionchetti P, Eliakim R, Ardizzone S, Armuzzi A, Barreiro-de Acosta M, Burisch J, Gecse KB, Hart AL, Hindryckx P, Langner C, Limdi JK, Pellino G, Zagorowicz E, Raine T, Harbord M, Rieder F; European Crohn's and Colitis Organisation [ECCO]. Third European Evidence-based Consensus on Diagnosis and Management of Ulcerative Colitis. Part 1: Definitions, Diagnosis, Extra-intestinal Manifestations, Pregnancy, Cancer Surveillance, Surgery, and Ileo-anal Pouch Disorders. J Crohns Colitis. 2017 Jun 1;11(6):649-670. doi: 10.1093/ecco-jcc/jjx008. No abstract available. PMID 28158501
- [Result] Tontini GE, Vecchi M, Pastorelli L, Neurath MF, Neumann H. Differential diagnosis in inflammatory bowel disease colitis: state of the art and future perspectives. World J Gastroenterol. 2015 Jan 7;21(1):21-46. doi: 10.3748/wjg.v21.i1.21. PMID 25574078
- [Result] Cartana ET, Gheonea DI, Saftoiu A. Advances in endoscopic ultrasound imaging of colorectal diseases. World J Gastroenterol. 2016 Feb 7;22(5):1756-66. doi: 10.3748/wjg.v22.i5.1756. PMID 26855535
- [Result] Ellrichmann M, Wietzke-Braun P, Dhar S, Nikolaus S, Arlt A, Bethge J, Kuehbacher T, Wintermeyer L, Balschun K, Klapper W, Schreiber S, Fritscher-Ravens A. Endoscopic ultrasound of the colon for the differentiation of Crohn's disease and ulcerative colitis in comparison with healthy controls. Aliment Pharmacol Ther. 2014 Apr;39(8):823-33. doi: 10.1111/apt.12671. Epub 2014 Feb 25. PMID 24612000
- [Derived] Nguyen VQ, Celio F, Chitnavis M, Shakhatreh M, Katz J, Cominelli F, Chak A, Yeaton P. Role of through-the-scope catheter-based EUS in inflammatory bowel disease diagnosis and activity assessment. Gastrointest Endosc. 2023 Apr;97(4):752-758.e2. doi: 10.1016/j.gie.2022.10.043. Epub 2022 Nov 4. PMID 36343674